CLINICAL TRIAL: NCT05887115
Title: Trial of Nurse Family Partnership for Women With Previous Live Births
Brief Title: Nurse Family Partnership for Women With Previous Live Births
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment milestones not met; funding withdrawn
Sponsor: University of Colorado, Denver (Other)
Collaborators: Nationwide Children's Hospital (Other); University of Rochester (Other); Columbia University (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-0470
Record Dates: First submitted 2023-04-27; First posted 2023-06-02 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy, High Risk; Child Development; Post Partum Depression
Keywords: Nurse Family Partnership; Home Visiting
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Research assistants will not collect any NFP program data - only equivalent research data in both control and NFP groups. Research assistants will remind participants not to tell the researchers which group they are in prior to each research data collection. We will also record in our participant tracking database if a researcher is ever "unmasked" (e.g., saw the NFP folder/ materials/participant mentioned their NFP nurse during an interview). Similarly, the nurses providing NFP will not be aware of which of their clients are involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (NFP) (Active Comparator): In the standard NFP intervention, low-income pregnant women are recruited to voluntarily join the program through their 28th week of pregnancy. Enrolled women receive home visits from a nurse. The visits can occur in-person or via telehealth. In-person visits can occur in the client's home or in another community location agreed upon by the client and the nurse (such as a library or coffee shop). The typical schedule for visits is weekly during the first month after enrollment, every two weeks until the birth of the infant, weekly during the post-partum period, then every two to four weeks until child age two.
  Interventions: Behavioral: Nurse Family Partnership
- Control (No Intervention): The control group will receive usual care for pregnant people, which may include home visiting services from another source other than NFP. Participants who are randomly selected to receive other services will be given information about other services for which they may qualify and information about how to access those services.

INTERVENTIONS:
Behavioral: Nurse Family Partnership — During NFP visits, the nurse: 1) engages in a therapeutic nurse-client relationship focused on promoting client abilities and behavior change to protect and promote her own health and child's health; 2) provides service coordination based on client's identified needs, referring to available community services; 3) follows NFP Visit Guidelines tailoring them to the strengths and challenges of each family; 4) works with client to support a healthy pregnancy by recognizing and reducing risk factors and promoting prenatal health care, healthy diet, exercise, and stress management; and 5) gathers data on program implementation and maternal and child health. The visits include content from six domains: personal health, environmental health, life-course, maternal role, family and friends, and health and human services. Nurses use educational materials to address the content from the six domains with their clients.
  Arms: Intervention (NFP)

SUMMARY:
The goal of this clinical trial is to test the Nurse Family Partnership (NFP) in mothers with previous live births (multiparous or multip individuals). The main aims are:

Specific Aim 1-Determine the effectiveness of NFP among multiparous women for reducing maternal morbidity and improving pregnancy outcomes.

Specific Aim 2-Determine the effectiveness of NFP among index children (child from pregnancy when mother was enrolled) of multiparous women for improving child outcomes.

Specific Aim 3 (Exploratory)-In preparation for a future study of the effects of preventive home-visiting programs on mother-index child-sibling triads, describe siblings (characteristics, role, influence) in the context of nurse home-visiting and evaluate the effectiveness of NFP on outcomes for prior-born siblings younger than 6 years old living in the home, including cognitive development, socioemotional development, and identification and referral to needed services.

A supplemental study to this study, led by investigators at Yale and Columbia, includes the following Aims:

Aim 1: Test whether the NFP causes variation in DNAm at Glucocorticoid-sensitive sites in infants over the first year of life.

Aim 2: Determine whether NFP causes differences in epigenetic age in infants over the first year of life.

Aim 3: Evaluate DNAm signatures as predictors of infant development at 12 months of age.

DETAILED DESCRIPTION:
The proposed study will be conducted in partnership with two or more NFP sites in Columbus and Dayton, Ohio. Investigators will work with pregnancy resource referral centers to identify a process that fits into each site's flow for identifying and recruiting eligible multiparous pregnant women at 32 weeks EGA (estimated gestational age) or less to participate in the study. The study will recruit 500 women to participate. Half will be receiving NFP and half will be receiving any other community services available outside of NFP. Researchers will compare the intervention group with the control group to test the effects described in the Aims above (as outlined in the following hypotheses).

Hypothesis 1-Compared to multiparous women who receive usual care, women who receive NFP will have reductions in pregnancy-related hypertension and tobacco use.

Hypothesis 2-Compared to children of women who receive usual care, those whose mothers receive NFP will have improved language development.

Supplemental study hypotheses:

Hypothesis 1: maternal NFP participation causes DNAm variation at glucocorticoid-sensitive sites across the genome at birth, controlling for genetic ancestry

Hypothesis 2: NFP participation reduces DNAm age acceleration from birth to 12 months of age, controlling for genetic variation.

Hypothesis 3: Glucocorticoid-sensitive DNAm and epigenetic aging in offspring measured across infancy (birth to 12 months) will correlate with infant development at 12 months.

Women will be asked to participate in four data collection episodes at study enrollment/baseline (prior to 36 weeks gestation), 6 to 8 weeks postpartum, and child ages 6 and 9 months, and (if consented), to an additional visit at child age 12 months for the supplemental DNAm study.

Researchers will use the following data sources for this study: 1) data routinely collected by the NFP team to determine enrollment and engagement in the NFP program of study participants randomized to NFP; 2) self-administered and interview surveys of study participants collected by the research assistant; 3) formal observation-based assessment tools (such as the Bayley assessment of child development) administered by the research assistant; 4) videos of parent-child interactions recorded by the research assistant and coded by parenting experts; 5) data from medical record review of mothers and their children; 6) birth certificate data; 7) buccal cell samples (infants) collected by the research assistant or self-collected by the participant with guidance from the research assistant.

The research assistants will conduct all the primary data collection from mother-child dyads who have agreed to participate in the trial, and primary data collection will be separate from NFP program delivery which will be conducted by the NFP nurses. Primary data collection will occur at 4 time points as described above. Primary data collection will occur in the participants' homes or at another location where the participant and research assistant feel comfortable (such as a meeting room in a public library). The majority of measures could be collected in a variety of settings with the exception of the video-taped interactions between parents and children which would ideally occur in the child's natural environment. The post partum and 6 month visits only involve maternal report measures and can be conducted by telephone/video using online surveys, unless the participant consents to the cheek swab at the post partum visit, which would be collected in-person.

The research assistant will record where each data collection episode occurred. The research assistant will also record all attempts made to contact study participants for data collection and missed episodes of data collection (i.e., if a visit were arranged and the participant were not available). The research assistant will be trained regarding appropriate collection, transport, and storage procedures for biologic samples and will be trained to conduct the Bayley assessment of child development.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant at 32 weeks EGA or less
2. history of previous live birth
3. covered by Medicaid or Medicaid-eligible
4. at least one of the following risks or adversities -age 19 or younger, no high school degree or equivalent, homeless (using a standardized definition), previous birth with low birth weight or prematurity, previous pregnancy with severe morbidity based on Centers for Disease Control definition, current pregnancy within 18 months of previous pregnancy, currently using tobacco or marijuana, history of substance use disorder, and self-identification as Black/African American (as a marker of facing the adversity of structural racism).

Exclusion Criteria:

1. unable converse and demonstrate adequate understanding to provide consent for study participation in English or Spanish
2. are already enrolled in a home-visiting intervention with this pregnancy
3. have previously been enrolled in NFP
4. under the age of 16 years. Note that we propose to exclude those who don't speak English or Spanish from our study because the community served by the two NFP delivery sites participating in our study is mostly English-speaking with some Spanish-speaking. However, those who don't speak English or Spanish are not excluded from participation in NFP, and NFP routinely provides services to all eligible families regardless of language spoken using bilingual/multilingual nurses when available or using interpretation services. NFP materials for nurses to use with families, known as 'facilitators', are available in several languages. In the rare circumstance that a pregnant woman is excluded from participating in our study based on language, they will not be excluded from receiving NFP.

Ages: 16 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participant must be pregnant to participate; can identify as any gender
Enrollment: 23 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Presence of Pregnancy-related hypertension | Birth of index child
  High Blood Pressure associated with pregnancy
Change in maternal tobacco use by cotinine | Less than 28 weeks gestation and 36 weeks gestation
  Measured by cotinine level in saliva
Change in self reported maternal tobacco use | Less than 36 weeks gestation, within 6 weeks of index birth (postpartum), index child age 6 months, 9 months
  Measured by self-report (yes/no)
Index child language development measured by the Bayley IV language subscale | Index child age 12 months
  Scaled, age-adjusted score from 1-19 with 19 being best outcome
Index child language development measured by the Peabody Picture Vocabulary Test | Index child age 9 months
  Percentage out of 100; 100 being best outcome
DNA methylation biomarkers | Within 6 weeks of index birth (postpartum) and child age 12 months
  Epigenetic age and glucocorticoid-sensitive DNA methylation score from methylation array data

SECONDARY OUTCOMES:
Number of participants with infection during pregnancy based on medical record review | Index child age 1 month
  Receipt of screening for common infections; if positive, receipt of appropriate treatment
Number of infants born with weight less than 2500 grams per medical record review | Index child age 1 month
Number of infants born less than 34 weeks gestation per medical record review | Index child age 1 month
Change in self-reported maternal substance use | Less than 36 weeks gestation, within 6 weeks of index birth (postpartum), index child age 6 months, 9 months
  Past month use per self-report (yes/no)
Initiation and continuation of any breastfeeding per maternal report | Index child age 1 month, 6 months
  Maternal report of any breastfeeding
Percentage of well-child visits attended for index child per medical record review | Index child age 9-12 months
  Number out of 6 visits by 9 months
Index child immunization use per medical record review | Record review at index child age 9-12 months
  Immunizations up-to-date for age at 9 months
Index child emergency room visits for serious preventable injuries and sentinel injuries for child abuse. | Index child age birth to 9 months, Record review at index child age 9-12 months
  Visit rate and reason for visit per medical record review
Index child hospitalization for injuries | Record review at index child age 9-12 months
  Number of days hospitalized for injury per medical record review
Change in quality of home environment measured by the HOME (Home Observation Measurement of the Environment) Inventory short form | 36 weeks gestation, index child age 6 months
  53 yes/no measures; score scaled based on child age, self-report and interviewer observation
Change in quality of home environment measured by the CHAOS (Confusion, Hubbub and Order Scale) Scale | 36 weeks gestation, index child age 6 months
  On a scale of 1-15, The higher the score the higher the level of environmental chaos in the home
Mother-child interaction measured by the Dyadic Assessment of Naturalistic Caregiver-child Experiences (DANCE) | Index child age 9 months
  Video recorded interactions are scored by trained research assistants, for each behavior the frequency and proportion of time spent is recorded.
Child's developmental index measured by Bayley IV developmental assessment | Index child age 12 months
  Scaled, age-adjusted score from 1-19 with 19 being best outcome
Index child's social and emotional development based on Bayley IV socio-emotional subscale | Index child age 12 months
  Scaled, age-adjusted score from 1-19 with 19 being best outcome
Index child's social and emotional development measured by the Child Behavior Checklist (CBCL) (maternal report) | Index child age 6 months
  54 question scored on a scale of 0-2; lower scores are more emotionally regulated children
Change in maternal perceived stress measured by Perceived Stress Scale (maternal report) | Less than 36 weeks gestation and index child age 6 months
  Scale of 0-40 based on 10 questions; 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy A Allison, MD, MSPH, Principal Investigator — University of Colorado School of Medicine; Deena Chisolm, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data with researchers who desire to conduct additional analyses. Investigators who are interested in accessing de-identified individual participant data should e-mail the Prevention Research Center for Family and Child Health (FamilyChildPRC@cuanschutz.edu) to request an application for data use. The leadership team at the PRC (Prevention Research Center for Family and Child Health) will review the application and determine whether to grant access. The criteria are listed below under 'Access Criteria'.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the close of currently funded study (January 2027) and will be available for 10 years (through December 2036).
Access Criteria: Criteria used in the review are as follows:
  1. Proposal has reasonable scientific merit; allows data to be put to good scientific use. Proposal is both theoretically and empirically sound.
     1. Statistical power is appropriate given level of project
     2. Likely usefulness for investigator.
     3. Likely to contribute to existing knowledge base
  2. Investigator's collaborator should be associated with our team. They provide link to our team, may provide access to data or at least communicate what data are available.
  3. Proposed analyses have not already been completed or proposed by other collaborators or members of the research team.
  4. Demands on current staff time are minimal including:
     1. Variable construction
     2. Statistical consultation
     3. Providing computer access/resources
     4. Data cleaning
     5. Providing access to data
     6. Current load of staff, including existing outside projects

REFERENCES:
- [Background] Bor J, Cohen GH, Galea S. Population health in an era of rising income inequality: USA, 1980-2015. Lancet. 2017 Apr 8;389(10077):1475-1490. doi: 10.1016/S0140-6736(17)30571-8. PMID 28402829
- [Background] Freudenberg N, Ruglis J. Reframing school dropout as a public health issue. Prev Chronic Dis. 2007 Oct;4(4):A107. Epub 2007 Sep 15. PMID 17875251
- [Background] Petersen EE, Davis NL, Goodman D, Cox S, Mayes N, Johnston E, Syverson C, Seed K, Shapiro-Mendoza CK, Callaghan WM, Barfield W. Vital Signs: Pregnancy-Related Deaths, United States, 2011-2015, and Strategies for Prevention, 13 States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2019 May 10;68(18):423-429. doi: 10.15585/mmwr.mm6818e1. PMID 31071074
- [Background] Wang E, Glazer KB, Howell EA, Janevic TM. Social Determinants of Pregnancy-Related Mortality and Morbidity in the United States: A Systematic Review. Obstet Gynecol. 2020 Apr;135(4):896-915. doi: 10.1097/AOG.0000000000003762. PMID 32168209
- [Background] Cheng TL, Johnson SB, Goodman E. Breaking the Intergenerational Cycle of Disadvantage: The Three Generation Approach. Pediatrics. 2016 Jun;137(6):e20152467. doi: 10.1542/peds.2015-2467. Epub 2016 May 9. PMID 27244844
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on Integrating the Science of Early Childhood Development; Shonkoff JP, Phillips DA, editors. From Neurons to Neighborhoods: The Science of Early Childhood Development. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225557/ PMID 25077268
- [Background] Noble KG, Houston SM, Brito NH, Bartsch H, Kan E, Kuperman JM, Akshoomoff N, Amaral DG, Bloss CS, Libiger O, Schork NJ, Murray SS, Casey BJ, Chang L, Ernst TM, Frazier JA, Gruen JR, Kennedy DN, Van Zijl P, Mostofsky S, Kaufmann WE, Kenet T, Dale AM, Jernigan TL, Sowell ER. Family income, parental education and brain structure in children and adolescents. Nat Neurosci. 2015 May;18(5):773-8. doi: 10.1038/nn.3983. Epub 2015 Mar 30. PMID 25821911
- [Background] Noble KG, Engelhardt LE, Brito NH, Mack LJ, Nail EJ, Angal J, Barr R, Fifer WP, Elliott AJ; PASS Network. Socioeconomic disparities in neurocognitive development in the first two years of life. Dev Psychobiol. 2015 Jul;57(5):535-51. doi: 10.1002/dev.21303. Epub 2015 Mar 30. PMID 25828052
- [Background] Brito NH, Noble KG. Socioeconomic status and structural brain development. Front Neurosci. 2014 Sep 4;8:276. doi: 10.3389/fnins.2014.00276. eCollection 2014. PMID 25249931
- [Background] Bradley RH, Corwyn RF. Socioeconomic status and child development. Annu Rev Psychol. 2002;53:371-99. doi: 10.1146/annurev.psych.53.100901.135233. PMID 11752490
- [Background] Duncan GJ, Dowsett CJ, Claessens A, Magnuson K, Huston AC, Klebanov P, Pagani LS, Feinstein L, Engel M, Brooks-Gunn J, Sexton H, Duckworth K, Japel C. School readiness and later achievement. Dev Psychol. 2007 Nov;43(6):1428-1446. doi: 10.1037/0012-1649.43.6.1428. PMID 18020822
- [Background] Uchino BN. Social support and health: a review of physiological processes potentially underlying links to disease outcomes. J Behav Med. 2006 Aug;29(4):377-87. doi: 10.1007/s10865-006-9056-5. Epub 2006 Jun 7. PMID 16758315
- [Background] Falk-Rafael A. Advancing nursing theory through theory-guided practice: the emergence of a critical caring perspective. ANS Adv Nurs Sci. 2005 Jan-Mar;28(1):38-49. doi: 10.1097/00012272-200501000-00005. PMID 15718937
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R, Chamberlin R. Improving the delivery of prenatal care and outcomes of pregnancy: a randomized trial of nurse home visitation. Pediatrics. 1986 Jan;77(1):16-28. PMID 3510017
- [Background] Olds DL, Henderson CR Jr, Chamberlin R, Tatelbaum R. Preventing child abuse and neglect: a randomized trial of nurse home visitation. Pediatrics. 1986 Jul;78(1):65-78. PMID 2425334
- [Background] Olds DL, Henderson CR Jr, Tatelbaum R, Chamberlin R. Improving the life-course development of socially disadvantaged mothers: a randomized trial of nurse home visitation. Am J Public Health. 1988 Nov;78(11):1436-45. doi: 10.2105/ajph.78.11.1436. PMID 3052116
- [Background] Olds DL, Eckenrode J, Henderson CR Jr, Kitzman H, Powers J, Cole R, Sidora K, Morris P, Pettitt LM, Luckey D. Long-term effects of home visitation on maternal life course and child abuse and neglect. Fifteen-year follow-up of a randomized trial. JAMA. 1997 Aug 27;278(8):637-43. PMID 9272895
- [Background] Olds D, Henderson CR Jr, Cole R, Eckenrode J, Kitzman H, Luckey D, Pettitt L, Sidora K, Morris P, Powers J. Long-term effects of nurse home visitation on children's criminal and antisocial behavior: 15-year follow-up of a randomized controlled trial. JAMA. 1998 Oct 14;280(14):1238-44. doi: 10.1001/jama.280.14.1238. PMID 9786373
- [Background] Kitzman H, Olds DL, Henderson CR Jr, Hanks C, Cole R, Tatelbaum R, McConnochie KM, Sidora K, Luckey DW, Shaver D, Engelhardt K, James D, Barnard K. Effect of prenatal and infancy home visitation by nurses on pregnancy outcomes, childhood injuries, and repeated childbearing. A randomized controlled trial. JAMA. 1997 Aug 27;278(8):644-52. PMID 9272896
- [Background] Kitzman H, Olds DL, Sidora K, Henderson CR Jr, Hanks C, Cole R, Luckey DW, Bondy J, Cole K, Glazner J. Enduring effects of nurse home visitation on maternal life course: a 3-year follow-up of a randomized trial. JAMA. 2000 Apr 19;283(15):1983-9. doi: 10.1001/jama.283.15.1983. PMID 10789666
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614
- [Background] Olds DL, Kitzman H, Hanks C, Cole R, Anson E, Sidora-Arcoleo K, Luckey DW, Henderson CR Jr, Holmberg J, Tutt RA, Stevenson AJ, Bondy J. Effects of nurse home visiting on maternal and child functioning: age-9 follow-up of a randomized trial. Pediatrics. 2007 Oct;120(4):e832-45. doi: 10.1542/peds.2006-2111. PMID 17908740
- [Background] Olds DL, Kitzman HJ, Cole RE, Hanks CA, Arcoleo KJ, Anson EA, Luckey DW, Knudtson MD, Henderson CR Jr, Bondy J, Stevenson AJ. Enduring effects of prenatal and infancy home visiting by nurses on maternal life course and government spending: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):419-24. doi: 10.1001/archpediatrics.2010.49. PMID 20439792
- [Background] Olds DL, Robinson J, O'Brien R, Luckey DW, Pettitt LM, Henderson CR Jr, Ng RK, Sheff KL, Korfmacher J, Hiatt S, Talmi A. Home visiting by paraprofessionals and by nurses: a randomized, controlled trial. Pediatrics. 2002 Sep;110(3):486-96. doi: 10.1542/peds.110.3.486. PMID 12205249
- [Background] Olds DL, Robinson J, Pettitt L, Luckey DW, Holmberg J, Ng RK, Isacks K, Sheff K, Henderson CR Jr. Effects of home visits by paraprofessionals and by nurses: age 4 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1560-8. doi: 10.1542/peds.2004-0961. PMID 15574615
- [Background] Olds DL, Holmberg JR, Donelan-McCall N, Luckey DW, Knudtson MD, Robinson J. Effects of home visits by paraprofessionals and by nurses on children: follow-up of a randomized trial at ages 6 and 9 years. JAMA Pediatr. 2014 Feb;168(2):114-21. doi: 10.1001/jamapediatrics.2013.3817. PMID 24296904
- [Background] Fraser JA, Armstrong KL, Morris JP, Dadds MR. Home visiting intervention for vulnerable families with newborns: follow-up results of a randomized controlled trial. Child Abuse Negl. 2000 Nov;24(11):1399-429. doi: 10.1016/s0145-2134(00)00193-9. PMID 11128173
- [Background] Alonso-Marsden S, Dodge KA, O'Donnell KJ, Murphy RA, Sato JM, Christopoulos C. Family risk as a predictor of initial engagement and follow-through in a universal nurse home visiting program to prevent child maltreatment. Child Abuse Negl. 2013 Aug;37(8):555-65. doi: 10.1016/j.chiabu.2013.03.012. Epub 2013 May 6. PMID 23660409
- [Background] Duggan A, Caldera D, Rodriguez K, Burrell L, Rohde C, Crowne SS. Impact of a statewide home visiting program to prevent child abuse. Child Abuse Negl. 2007 Aug;31(8):801-27. doi: 10.1016/j.chiabu.2006.06.011. Epub 2007 Sep 5. PMID 17822764
- [Background] DuMont K, Mitchell-Herzfeld S, Greene R, Lee E, Lowenfels A, Rodriguez M, Dorabawila V. Healthy Families New York (HFNY) randomized trial: effects on early child abuse and neglect. Child Abuse Negl. 2008 Mar;32(3):295-315. doi: 10.1016/j.chiabu.2007.07.007. PMID 18377991
- [Background] Bowlby J. Attachment and loss: retrospect and prospect. Am J Orthopsychiatry. 1982 Oct;52(4):664-678. doi: 10.1111/j.1939-0025.1982.tb01456.x. No abstract available. PMID 7148988
- [Background] Swain JE, Kim P, Spicer J, Ho SS, Dayton CJ, Elmadih A, Abel KM. Approaching the biology of human parental attachment: brain imaging, oxytocin and coordinated assessments of mothers and fathers. Brain Res. 2014 Sep 11;1580:78-101. doi: 10.1016/j.brainres.2014.03.007. Epub 2014 Mar 15. PMID 24637261
- [Background] Evans GW, Gonnella C, Marcynyszyn LA, Gentile L, Salpekar N. The role of chaos in poverty and children's socioemotional adjustment. Psychol Sci. 2005 Jul;16(7):560-5. doi: 10.1111/j.0956-7976.2005.01575.x. PMID 16008790
- [Background] Miller TR. Projected Outcomes of Nurse-Family Partnership Home Visitation During 1996-2013, USA. Prev Sci. 2015 Aug;16(6):765-77. doi: 10.1007/s11121-015-0572-9. PMID 26076883
- [Background] Bandura A. Self-efficacy: The exercise of control. Macmillan; 1997 Feb 15.
- [Background] Bandura A. Social foundations of thought and action. Englewood Cliffs, NJ. 1986;1986(23-28):2.
- [Background] Bronfenbrenner U. Toward an experimental ecology of human development. American psychologist. 1977;32(7):513.
- See also: Braveman PE, S. . Overcoming Obstacles to Health in 2013 and Beyond. RQJF Commission to Build a Healthier America https://www.rwjf.org/en/library/research/2013/06/overcoming-obstacles-to-health-in-2013-and-beyond.html. Published 2013. Accessed2019. — http://www.commissiononhealth.org/PDF/ObstaclesToHealth-Report.pdf
- See also: McIntosh K, Moss, E., Nunn, R., and Shambaugh, J. Examining the Black-white wealth gap. The Brookings Institute. https://www.brookings.edu/blog/up-front/2020/02/27/examining-the-black-white-wealth-gap/. Published 2020. Accessed2020. — https://www.brookings.edu/blog/up-front/2020/02/27/examining-the-black-white-wealth-gap/.
- See also: Darity Jr. W, Hamilton, D., Paul, M., Aja, A., Price, A., Moore, A., and Chiopris, C. What We Get Wrong About Closing the Racial Wealth Gap. Samuel DuBois Cook Center on Social Equality, Insight Center for Community Economic Development. — https://socialequity.duke.edu/wp-content/uploads/2019/10/what-we-get-wrong.pdf
- See also: Hart B, Risley TR. The early catastrophe. EDUCATION REVIEW-LONDON-. 2003;17(1):110-118. — https://www.aft.org/ae/spring2003/hart_risley
- See also: Nurse-Family Partnership: A nurse home visitation program for low-income, pregnant women. Social Programs that Work. Prenatal/Early Childhood. . https://evidencebasedprograms.org/policy_area/prenatal-earlychildhood/. Published 2019. Accessed 6/12/2019. — https://evidencebasedprograms.org/policy_area/prenatal-earlychildhood
- See also: Effectiveness HVEo. What is Home Visiting Evidence of Effectiveness? U.S. Department of Health and Human Serivces: Administration for Children and Families. https://homvee.acf.hhs.gov/. Published 2020. Accessed2020. — https://homvee.acf.hhs.gov/
- See also: Haskins R, Paxson, C., Brooks-Gunn, J. Social Science Rising: A Tale of Evidence Shaping Public Policy. Princeton, Brookings. ;2009. — https://www.brookings.edu/wp-content/uploads/2016/06/1001_social_science_haskins.pdf

DOCUMENTS (1):
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT05887115/ICF_001.pdf